CLINICAL TRIAL: NCT03417739
Title: A Phase II Study of BVD-523 in Metastatic Uveal Melanoma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: BioMed Valley Discoveries, Inc (Industry)
Responsible Party: Principal Investigator, Elizabeth Buchbinder, MD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17-526
Record Dates: First submitted 2018-01-25; First posted 2018-01-31 (Actual); Results first posted 2021-11-11 (Actual); Last update posted 2024-06-25 (Actual); Status verified 2024-06

CONDITIONS: Uveal Melanoma
Keywords: Uveal Melanoma
MeSH Terms: conditions — Uveal Melanoma | interventions — ulixertinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- BVD-523 (Experimental): BVD-523 is administered at the RP2D of 600mgs taken twice daily orally for 28 consecutive days (1 cycle). Planned does may modified based on toxicity.
  Interventions: Drug: BVD-523

INTERVENTIONS:
Drug: BVD-523 — ERK1 and ERK2 inhibitor
  Other Names: Ulixertinib

SUMMARY:
This research study is studying a targeted therapy called BVD-523 as a possible treatment for advanced uveal melanoma.

DETAILED DESCRIPTION:
This research study is a Phase II clinical trial. Phase II clinical trials test the safety and effectiveness of an investigational drug to learn whether the drug works in treating a specific disease. "Investigational" means that the drug is being studied.

The FDA (the U.S. Food and Drug Administration) has not approved BVD-523 as a treatment for any disease.

BVD-523 has been tested in patients with solid tumors to determine the highest dose of BVD-523 that can be safely given to patients.

In this research study, the investigators are evaluating the role of BVD-523 in the treatment of patients with uveal melanoma. Genetic changes within metastatic uveal melanoma activate proteins in the MAPK protein signaling pathway which leads to tumor growth. In the laboratory BVD-523 works against one of these proteins called ERK to decrease tumor growth. In this study, the investigators are testing BVD-523 to see if it works to treat metastatic uveal melanoma.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have histologically or cytologically confirmed stage IV uveal melanoma
* Participants must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded for non-nodal lesions and short axis for nodal lesions) as ≥20 mm with conventional techniques or as ≥10 mm with spiral CT scan, MRI, or calipers by clinical exam. See Section 11 for the evaluation of measurable disease.
* Patients can have received any number of prior therapies for treatment of their uveal melanoma excluding prior treatment with an ERK inhibitor. Patients who have received prior MEK inhibition or other MAPK targeted agents will be allowed on study.
* Age ≥ 18 years of age.
* ECOG performance status ≤2 (Karnofsky ≥60%, see Appendix A)
* Life expectancy of greater than 6 months
* Participants must have normal organ and marrow function as defined below:

  * leukocytes ≥3,000/mcL
  * hemoglobin ≥9.0 g/dL
  * absolute neutrophil count ≥1,500/mcL
  * platelets ≥100,000/mcL
  * total bilirubin ≤1.5 × institutional upper limit of normal AST(SGOT)/ALT(SGPT) ≤2.5 × institutional upper limit of normal, unless there is known liver involvement in which case ≤5.0 × institutional upper limit of normal
  * creatinine within normal institutional limits OR
  * creatinine clearance ≥60 mL/min/1.73 m2 for participants with creatinine levels above institutional normal.
* Participants must have adequate cardiac function, e.g. left ventricular ejection fraction (LVEF) of >50% as assessed by multi-gated acquisition (MUGA) or ultrasound/echocardiography (ECHO); corrected QT interval (QTc) <470ms.
* Presence of metastatic disease that would be amenable to the required biopsies. Ideally pre and post biopsies should be from the same lesion and otherwise from lesions in the same organ. If not possible, then biopsy of the lesions in different organs will be permitted.
* The effects of BVD-523 on the developing human fetus are unknown. For this reason and because ERK inhibitors could potentially be teratogenic, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and 4 months after completion of BVD-523 administration. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 4 months after completion of BVD-523 administration.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Participants who have had chemotherapy or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C), small molecule targeted therapy (i.e. - kinase inhibitors) within 3 weeks or the last dose of antibody therapy within 4 weeks prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier.
* Participants who are receiving any other investigational agents.
* Major surgery within 4 weeks of the first dose of BVD-523. Tumor embolization procedure or ablation procedure within 2 weeks of first dose of BVD-523.
* Participants with known brain metastases or evidence of leptomeningeal involvement are eligible only if these lesions are treated and both clinically and radiographically stable for at least four weeks. Patients are eligible if they are being treated with a stable dosage of steroids/anticonvulsants, requiring no dose increase for 4 weeks.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to BVD-523.
* Participants receiving any medications or substances that are known to be strong inhibitors of CYP1A2, CYP2D6, and CYP3A4 or strong inducers of CYP3A4 are ineligible. Because the lists of these agents are constantly changing, it is important to regularly consult a frequently-updated list such as http://medicine.iupui.edu/clinpharm/ddis/table.aspx; medical reference texts such as the Physicians' Desk Reference may also provide this information. As part of the enrollment/informed consent procedures, the patient will be counseled on the risk of interactions with other agents, and what to do if new medications need to be prescribed or if the patient is considering a new over-the-counter medicine or herbal product.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant women are excluded from this study because BVD-523 is an ERK with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with BVD-523 breastfeeding should be discontinued if the mother is treated with BVD-523.
* Gastrointestinal (GI) condition which could impair absorption of study medication or inability to ingest study medication.
* A history of current evidence/risk of retinal vein occlusion (RVO) or central serous retinopathy (CSR)
* Concomitant malignancies or previous malignancies with less than 2 years of disease-free interval at the time of enrollment (except non-melanoma skin cancer, cervical cancer in situ, prostate cancer with undetectable PSA). Other concurrent malignancies must be discussed with the medical monitor prior to enrollment.
* Patients with melanoma of cutaneous, mucosal or acral-lentiginous origin or of unknown primary.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2018-03-26 (Actual); Primary Completion 2020-05-05 (Actual); Study Completion 2025-08-31 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Buchbinder, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (2):
- United States (2):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | BVD-523
Started | 13
Completed | 13
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | BVD-523
Number analyzed (Participants) | 13
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.1 (10.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 4
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 1
  White | 12
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 13

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate
Description: Overall Response Rate (ORR) was defined as the proportion of participants achieving complete response (CR) or partial response (PR) based on RECIST 1.1 criteria on treatment. Per RECIST 1.1 for target lesions: CR is complete disappearance of all target lesions and PR is at least a 30% decrease in the sum of longest diameter (LD) of target lesions, taking as reference baseline sum LD. PR or better overall response assumes at a minimum incomplete response/stable disease (SD) for the evaluation of non-target lesions and absence of new lesions.
Time Frame: up to 52 weeks
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | BVD-523
Number analyzed (Participants) | 13
percentage of participants | 0 [0 to 20.5]

2. Secondary Outcome: Disease Control Rate
Description: A combination of patients who experience complete response, partial response and stable disease on CT or other form of imaging
Time Frame: up to 52 weeks
Measure: Number; unit: percentage of participants
Arm/Group | BVD-523
Number analyzed (Participants) | 13
percentage of participants | 0

3. Secondary Outcome: Median Overall Survival
Description: OS based on the Kaplan-Meier method is defined as the time from study entry to death or censored at date last known alive.
Time Frame: Participant survival information will be collected every 4 weeks from the date of last dose of study drug until the participant's death or until the participant is lost to follow-up, or until study closure. Median follow-up was 6 months.
Measure: Median (90% Confidence Interval); unit: Months
Arm/Group | BVD-523
Number analyzed (Participants) | 13
Months | 6.9 [3.2 to 8.3]

4. Secondary Outcome: Median Time to Tumor Progression
Description: Time from enrollment on study until the tumor is progressing by RECIST v1.0 as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions
Time Frame: Between the dates of the start of trial treatment and first documentation of progressive disease. In the absence of documented progressive disease, follow-up will be censored at date of last disease assessment. up to 52 weeks
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | BVD-523
Number analyzed (Participants) | 13
months | 2 [1.8 to 3.6]

5. Secondary Outcome: To Evaluate the Pharmacodynamics of ERK Inhibition on BVD-523 With a Comparison of Pre- and On-treatment Biopsies.
Description: MAPK pathway inhibition will be analyzed in pre-treatment and post-treatment samples to understand the effect of ERK inhibition by BVD-523
Time Frame: Tumor biopsies are obtained 7-28 days prior to the first treatment and 12-16 days following the initial treatment in order to facilitate ERK signaling analysis, mutation analysis, sequencing, and cell line development.
Reporting Status: Not Posted, anticipated posting 2024-12

6. Secondary Outcome: To Better Understand the Genetic Variability of Uveal Melanoma Through Whole Exome Sequencing
Description: DNA sequencing will occur in tissue samples from patients treated on study to gain a better understanding of the genetic variability observed in uveal melanoma
Time Frame: as for outcome 5
Reporting Status: Not Posted, anticipated posting 2024-12

ADVERSE EVENTS:
Time Frame: AE data collected at day 1 of each cycle, and day 15 of cycle 1, days 22 to 28 of cycle 2. Also during off treatment follow-up. AE will be collected every 4 weeks from the date of last dose of study drug until the participant's death or until the participant is lost to follow-up, or until study closure up to one year.
Description: Serious AEs (SAE) were defined as events with treatment-attribution of possibly, probably or definitely and grade 3 or higher. All remaining AEs are classified as Other AEs (OAE) including grade 3 or higher events with treatment-attribution of unlikely and unrelated plus all grade 1 and 2 events. Maximum grade toxicity by type was then calculated within SAE and OAE datasets. No further data is available to specify classification of other beyond the general term.
Arm/Group | BVD-523
All-Cause Mortality (participants affected / at risk) | 0/13
Serious Adverse Events (participants affected / at risk) | 5/13
Other Adverse Events (participants affected / at risk) | 13/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | BVD-523 (N=13)
Anemia (Blood and lymphatic system disorders) | 1
Alanine aminotransferase increased (Investigations) | 2
Aspartate aminotransferase increased (Investigations) | 2
Serum amylase increased (Investigations) | 1
Hyponatremia (Metabolism and nutrition disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | BVD-523 (N=13)
Anemia (Blood and lymphatic system disorders) | 1
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 1
Lymph node pain (Blood and lymphatic system disorders) | 1
Palpitations (Cardiac disorders) | 1
Supraventricular tachycardia (Cardiac disorders) | 1
Blurred vision (Eye disorders) | 1
Eye disorders - Other, specify (Eye disorders) | 2
Abdominal distension (Gastrointestinal disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 6
Anal ulcer (Gastrointestinal disorders) | 1
Ascites (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 3
Diarrhea (Gastrointestinal disorders) | 10
Esophageal stenosis (Gastrointestinal disorders) | 1
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 3
Gingival pain (Gastrointestinal disorders) | 1
Hemorrhoids (Gastrointestinal disorders) | 1
Mucositis oral (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 8
Rectal ulcer (Gastrointestinal disorders) | 1
Stomach pain (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 2
Chills (General disorders) | 1
Edema limbs (General disorders) | 4
Fatigue (General disorders) | 7
Fever (General disorders) | 3
Gait disturbance (General disorders) | 1
General disorders and administration site conditions - Other, specify (General disorders) | 3
Non-cardiac chest pain (General disorders) | 1
Pain (General disorders) | 1
Urinary tract infection (Infections and infestations) | 1
Bruising (Injury, poisoning and procedural complications) | 1
Fracture (Injury, poisoning and procedural complications) | 2
Alanine aminotransferase increased (Investigations) | 2
Alkaline phosphatase increased (Investigations) | 1
Aspartate aminotransferase increased (Investigations) | 2
Blood bilirubin increased (Investigations) | 1
CPK increased (Investigations) | 1
Creatinine increased (Investigations) | 3
Platelet count decreased (Investigations) | 1
Serum amylase increased (Investigations) | 1
Weight loss (Investigations) | 1
White blood cell decreased (Investigations) | 1
Anorexia (Metabolism and nutrition disorders) | 7
Dehydration (Metabolism and nutrition disorders) | 3
Hypoalbuminemia (Metabolism and nutrition disorders) | 4
Hypocalcemia (Metabolism and nutrition disorders) | 1
Hypokalemia (Metabolism and nutrition disorders) | 1
Hypomagnesemia (Metabolism and nutrition disorders) | 1
Hyponatremia (Metabolism and nutrition disorders) | 2
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Dizziness (Nervous system disorders) | 3
Dysgeusia (Nervous system disorders) | 1
Tremor (Nervous system disorders) | 1
Agitation (Psychiatric disorders) | 1
Anxiety (Psychiatric disorders) | 2
Confusion (Psychiatric disorders) | 1
Depression (Psychiatric disorders) | 1
Hematuria (Renal and urinary disorders) | 3
Urine discoloration (Renal and urinary disorders) | 1
Vaginal inflammation (Reproductive system and breast disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 3
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 2
Dry skin (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 5
Rash acneiform (Skin and subcutaneous tissue disorders) | 7
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 4
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 3
Hot flashes (Vascular disorders) | 1
Hypotension (Vascular disorders) | 2
Thromboembolic event (Vascular disorders) | 1
Vascular disorders - Other, specify (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-01-23): https://cdn.clinicaltrials.gov/large-docs/39/NCT03417739/Prot_SAP_000.pdf